CLINICAL TRIAL: NCT00815100
Title: Randomised, Double-blind, Placebo-controlled Trial of IVabradine in Patients With Acute Coronary Syndrome: Effects of the If Current Inhibitor Ivabradine or rEduction of Inflammation maRkers in Patients With Acute Coronary Syndrome
Brief Title: Effects of the Ivabradine on Reduction of Inflammatory Markers in Patients With Acute Coronary Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario de Canarias (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Riviera/09
Record Dates: First submitted 2008-12-25; First posted 2008-12-29 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Acute Coronary Syndromes
Keywords: Ivabradine; Acute coronary syndrome.; Inflammation; C-reactive protein; Atherosclerosis
MeSH Terms: conditions — Acute Coronary Syndrome; Inflammation; Atherosclerosis | interventions — Ivabradine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Ivabradine (Active Comparator)
  Interventions: Drug: Ivabradine

INTERVENTIONS:
Drug: Ivabradine — Eligible patients will be randomized to 1 of the 2 treatment arms, namely, double-blind ivabradine, or placebo, after hospital admission (at 48 hours). The starting dose of ivabradine will be 5 mg (or matching placebo) twice daily in all patients. Patients receiving 5 mg twice daily (or matching placebo) 1 week after the inclusion with a resting HR of ≥60 beats per minute will receive the target dose of 7.5 mg twice daily (or matching placebo).
  Arms: Ivabradine
Drug: Placebo — Eligible patients will be randomized to 1 of the 2 treatment arms, namely, double-blind ivabradine, or placebo, after hospital admission (at 48 hours). The starting dose of ivabradine will be 5 mg (or matching placebo) twice daily in all patients. Patients receiving 5 mg twice daily (or matching placebo) 1 week after the inclusion with a resting HR of ≥60 beats per minute will receive the target dose of 7.5 mg twice daily (or matching placebo).
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate whether a pure heart rate-lowering agent (Ivabradine) reduces vascular inflammatory stress in patients with acute coronary syndromes

DETAILED DESCRIPTION:
The activation of inflammatory pathways plays an important contributory role in coronary plaque instability and subsequent rupture, which can lead to the development of acute coronary syndromes. Elevated levels of serum inflammatory markers such as high-sensitivity C-reactive protein (hs-CRP) represent independent risk factors for further cardiovascular events. Raised resting heart rate (HR) has been shown to be associated with cardiovascular events. Ivabradine is a new HR-reducing agent, which has demonstrated antianginal and anti-ischemic properties in patients with stable angina. In an atherosclerosis model, selective HR reduction with ivabradine has been shown to decrease markers of vascular oxidative stress, to improve endothelial function, and to reduce atherosclerotic plaque formation. We hypothesized that the addition of ivabradine to standard medical therapy has a beneficial effect on markers of inflammatory stress in acute coronary syndrome patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female.
2. Age > 18 years.
3. Ischemic symptoms suspected to represent a non-ST segment elevation acute coronary syndrome defined as:

   Clinical history consistent with new onset, or a worsening pattern, of characteristic ischemic chest pain occuring at rest or with minimal exertion (lasting longer than 10 min) and planned to be managed with an early invasive strategy with intention to perform a percutaneous coronary intervention as early as possible and not later than 72 hours of randomization, and at least one of the following:
   1. ECG changes compatible with new ischemia (ST depression of at least 1 mm or transient ST elevation or ST elevation of <1 mm or T wave inversion >3 mm in at least 2 contiguous leads; or
   2. Already elevated cardiac enzymes (eg, CK-MB) or biomarkers (troponin I or T) above the upper limit of normal.
4. Patients should be in sinus rhythm with a resting HR of > 60 beats per minute on a resting standard 12-lead ECG.
5. Written informed consent obtained.

Exclusion Criteria:

1. Patients unlikely to cooperate in the study or with inability or unwillingness to give informed consent.
2. Pregnant or breast-feeding women or women of childbearing potential.
3. Patients with recent (< 6 months) myocardial infarction or coronary revascularization or with a history of stroke or cerebral transient ischemic attack within the preceding 3 months or scheduled for revascularization (percutaneous coronary intervention and coronary artery bypass graft).
4. Patients with at least 1 of the following criteria:

   * Implanted pacemaker or implantable cardioverter defibrillator.
   * Valvular disease likely to require surgery within the next 2 years.
   * Sick sinus syndrome, sinoatrial block, congenital long QT syndrome, complete atrioventricular block.
   * Expectation of death from other illness during the course of the trial.
   * Known severe liver or renal disease.
   * Requiring or likely to require the following medications: macrolide antibiotics, cyclosporin, gestodene, antiretroviral drugs or azole antifungals such as ketoconazole or with known hereditary problems of galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
5. Patients with systemic or cardiac inflammatory processes with the exception of atherosclerosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2011-09-07 (Actual)

PRIMARY OUTCOMES:
Whether initiation of ivabradine therapy in patients with acute coronary syndromes immediately after hospital admission decreases high-sensitivity C-reactive protein. | day 4 and day 30

SECONDARY OUTCOMES:
Whether initiation of ivabradine therapy decreases the occurrence of ischemic events (death, nonfatal myocardial infarction, unstable angina, urgent revascularization, cardiac arrest) in patients with acute coronary syndromes. | day 30, 90, 180 and 360

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife, Spain